CLINICAL TRIAL: NCT05299229
Title: Continuous Non-invasive Hemodynamic Monitoring in Early-onset Severe Preeclampsia: a Comparison of Echocardiography, Bioreactance, and Finger Cuff Measurements
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000028142
Record Dates: First submitted 2021-10-13; First posted 2022-03-28 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Heart and vascular function: All study participants will have echocardiography and non-invasive monitoring by chest/back sensors and a finger cuff to determine the best method of monitoring heart and vascular function in preeclampsia.
  Interventions: Diagnostic Test: Echocardiogrpahy and non-invasive monitoring

INTERVENTIONS:
Diagnostic Test: Echocardiogrpahy and non-invasive monitoring — Study participants will have echocardiography and non-invasive monitoring by chest/back sensors and a finger cuff.

SUMMARY:
The purpose of this study is to compare the feasibility and accuracy of two methods of non-invasive hemodynamic assessments - bioreactance as assessed by non-invasive cardiac output monitoring (NICOM; Cheetah Medical) and pulse wave analysis as assessed by finger cuff arterial pressure (ClearSite, Edwards Life Sciences) - compared to hemodynamic assessments by intermittent echocardiography in early onset preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* BP >160 or DBP >110
* gestational age between 20-34 weeks
* singleton pregnancy

Exclusion Criteria:

* prior diagnosis of chronic hypertension or hypertensive disorder of pregnancy
* multi-fetal pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with severe preeclampsia.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in cardiac output (L/min) as measured by NICOM (bioreactance) monitoring | Baseline (typically 3-5 days before birth, but can be up to 5 weeks before birth), 3 days after birth (postpartum)
  Cardiac output (L/min) ranges 3-10 L/min, lower values associated with more severe preeclampsia
Change in systemic vascular resistance (dynes/sec*cm-5) as measured by NICOM (bioreactance) monitoring | Baseline (typically 3-5 days before birth, but can be up to 5 weeks before birth), 3 days after birth (postpartum)
  Systemic vascular resistance ranges 600-2000 dynes/sec*cm-5, higher values associated with more severe preeclampsia
Change in Cardiac output (L/min) as measured by Clearsite (pulse wave analysis) monitoring | Baseline (typically 3-5 days before birth, but can be up to 5 weeks before birth), 3 days after birth (postpartum)
  Cardiac output (L/min) ranges 3-10 L/min, lower values associated with more severe preeclampsia
Change in Systemic vascular resistance (dynes/sec*cm-5) as measured by Clearsite (pulse wave analysis) monitoring | Baseline (typically 3-5 days before birth, but can be up to 5 weeks before birth), 3 days after birth (postpartum)
  Systemic vascular resistance ranges 600-2000 dynes/sec*cm-5, higher values associated with more severe preeclampsiaanalysis) monitoring
Change in Cardiac output (L/min) as measured by transthoracic echocardiography | Baseline (typically 3-5 days before birth, but can be up to 5 weeks before birth), 3 days after birth (postpartum)
  Cardiac output (L/min) ranges 3-10 L/min, lower values associated with more severe preeclampsia
Change in Systemic vascular resistance (dynes/sec*cm-5) as measured by transthoracic echocardiography | Baseline (typically 3-5 days before birth, but can be up to 5 weeks before birth), 3 days after birth (postpartum)
  Systemic vascular resistance ranges 600-2000 dynes/sec*cm-5, higher values associated with more severe preeclampsia

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No